CLINICAL TRIAL: NCT01695629
Title: In Vivo Corneal Confocal Microscopy for Non-invasive Assessment of Diabetic Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roni Shtein, Assistant Professor, Department of Ophthalmology, University of Michigan
Other Study IDs: DPN-42377
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin biopsy from leg
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- None to Mild: Subjects with Diabetes with none to mild peripheral neuropathy
- Severe: Subjects with diabetes with severe neuropathy

SUMMARY:
Clinical in vivo confocal microscopy (IVCM) is a relatively new technique of corneal evaluation that permits non-invasive imaging of corneal structures on the cellular level. Precise anatomic characterization of corneal structures, including corneal nerves, can be rapidly performed with high resolution.

DETAILED DESCRIPTION:
Evaluation of the corneal nerve layer with IVCM provides a method of direct visualization of peripheral small fiber nerves and a quantifiable assessment of nerve abnormalities in a low risk, non-invasive manner. Therefore, our goal is to develop a non-invasive diagnostic protocol as a quantitative tool for the evaluation of DPN. The protocol and the tool we seek to develop could ultimately be used in large-scale clinical trials and in clinical practice to assess DPN severity and progression.

We hypothesize that in vivo confocal imaging of the corneal nerve layer is a clinically viable method to assess and quantify systemic peripheral nerve health. We emphasize that this imaging method can be used in both humans and animal models to provide quantifiable, longitudinal data on the same live individual to advance our understanding of the development and progression of DPN, and to evaluate treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* diabetes

Exclusion Criteria:

* history of laser eye surgery, corneal disease, multiple sclerosis, Parkinson's disease, or any known systemic neuropathy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjes\cts with diabetes with none, mild or severe neuropathy
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
changes between control and diabetic patients | 12 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kellogg Eye Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] DeMill DL, Hussain M, Pop-Busui R, Shtein RM. Ocular surface disease in patients with diabetic peripheral neuropathy. Br J Ophthalmol. 2016 Jul;100(7):924-928. doi: 10.1136/bjophthalmol-2015-307369. Epub 2015 Oct 23. PMID 26500330